CLINICAL TRIAL: NCT03676777
Title: Prospective, Non-interventional, Multicenter Observational Study of Bacterial/Fungal Infections in Hospitalized Patients With Liver Cirrhosis in China
Brief Title: Study Of Bacterial/Fungal Infections in Hospitalized Patients With Liver Cirrhosis in China
Acronym: SONIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Qing XIe, Head of the Department of Infectious diseases, Ruijin Hospital, Ruijin Hospital
Other Study IDs: SONIC
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Cirrhosis
Keywords: Bacterial infection; Fungal infection; Cirrhosis; Multi-drug resistance; Antibiotic treatment; Clinical outcome; Organ failure; Acute-on-chronic liver failure; Decompensated cirrhosis; Complications of cirrhosis; Acute kidney injury
MeSH Terms: conditions — Fibrosis; Bacterial Infections; Mycoses; Acute-On-Chronic Liver Failure; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Serum; Plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infection: Patients admitted or developed bacterial/fungal infection while hospitalization
- Non-infection: Patients without bacterial/fungal infection

SUMMARY:
This is a national, investigator-initiated, multicenter, prospective, observational, web-based registry in hospitalized patients with cirrhosis across China.

The overarching aim of this study is to investigate the epidemiology and clinical impact of bacterial/fungal infections in hospitalized patients with liver cirrhosis in China within the collaborative network. We also aimed to build up the national prospective cohort of hospitalized cirrhosis in China to stand in the future for the backbone of various research programs focused on infection, other complications of cirrhosis, organ failure, the ACLF syndrome, end-stage liver disease and beyond.

DETAILED DESCRIPTION:
Patients with cirrhosis are prone to infections due to the abnormal bacterial translocation and immune dysfunction. Infections are more common when these patients are admitted into the hospital. Infections are life-threatening complications of cirrhosis which can precipitate hepatic encephalopathy, acute kidney injury, and the acute-on-chronic liver failure (ACLF) syndrome. The survival rate is significantly decreased once infections set in, especially when the first-line empirical antibiotic therapy is insufficient or inappropriate. Moreover, the prevalence of multi-drug-resistant organism (MDRO) is naturally increasing across the world due to the overuse of antibiotics. Patients with cirrhosis, especially those at the decompensated stage are at high risk of developing MDRO due to recurrent hospitalizations and repeatedly exposed to antibiotics either for treatment or prophylactic purposes. Empiric antibiotic therapy could be very difficult without understanding the profile of antibiotic resistance and could be varied significantly among different areas.

The issue of infection in patients with cirrhosis has been recently highlighted by International Club of Ascites with its "GLOBAL" study (ILC2018, GS-001) showing that the global prevalence of MDRO across the world was 34% (95% CI=31-37%). The prevalence of MDRO varies across the world with the highest in India followed by South America and other Asian countries. The source of acquisition (Community acquire, health-care related or nosocomial origin), site of infection (Spontaneous bacterial peritonitis, urinary tract, blood, respiratory tract, etc.) and category of the organism (Gram negative or positive) had an influence on the prevalence of MDRO and response to empirical antibiotic treatment. The results highlight the need to develop different empirical antibiotic strategies across different continents and countries, although China was not included in this study. Epidemiology data and investigation on the role of bacterial/fungal infection in patients with cirrhosis from China is therefore urgently needed.

The overarching aim of this study is to investigate the epidemiology and clinical impact of bacterial/fungal infections in hospitalized patients with liver cirrhosis in China within the collaborative network. We also aimed to build up the national prospective cohort of hospitalized cirrhosis in China to stand in the future for the backbone of various research programs focused on infection, other complications of cirrhosis, organ failure, the ACLF syndrome, end-stage liver disease and beyond.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient with cirrhosis as confirmed either by the histological scoring system, imaging technique (abdominal Ultrasound, CT or MRI), endoscopic findings or a combination of biochemical and clinical manifestation.
* Admitted for at least one of the following reasons:

  1. Bacterial infection/fungal infection
  2. Overt Ascites (Grade II-III)
  3. Gastrointestinal bleeding
  4. Hepatic encephalopathy
  5. Jaundice (Total bilirubin ≥5 mg/dL) with coagulation dysfunction (INR ≥1.5)

Exclusion Criteria:

* 1. Age below 16 or over 80 years
* 2. Lactation/ Pregnancy women
* 3. HIV infection
* 4. Admitted for scheduled procedures (e.g., band ligation, splenectomy, transjugular intrahepatic portosystemic shunting, liver biopsy) or re-examination or multidisciplinary consultation)
* 5. Hepatocellular carcinoma (HCC) outside Milan criteria or other disseminated malignancies
* 6. Previous liver transplantation
* 7. With previously known severe extra-hepatic diseases (e.g., chronic renal failure requiring hemodialysis, severe heart disease; severe chronic pulmonary disease, psychiatric disorders)
* 8. Taking immunosuppressive or anticoagulation drugs for the treatment of extra-hepatic disease.
* 9. Patient' s refusal to participation
* 10. Failure to provide prior informed consent or with documented evidence that the patient has no legal surrogate decision maker and it appears unlikely that the patient will regain consciousness or sufficient ability to provide delayed informed consent

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients with cirrhosis evaluated in a dedicated and organized tertiary-care center (Liver Unit, Department of infectious diseases, Department of Gastroenterology, emergency department) across China.
Sampling Method: Probability Sample
Enrollment: 1232 (Estimated)
Dates: Start 2018-11-07 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
28-day transplantation-free Survival | From admission to 28-day post-admission
  Survival at 28-day follow-up without liver transplantation

SECONDARY OUTCOMES:
Characteristics of bacterial/fungal infection including the prevalence of infection, the source of acquisition, type of infection, multidrug resistance rate, antibiotic treatment efficiency and efficacy in relation to disease course and outcome | From admission to discharge, an average of 28-day
  Characteristics of bacterial/fungal infection including the prevalence of infection, the source of acquisition, type of infection, multidrug resistance rate, antibiotic treatment efficiency and efficacy in relation to disease course and outcome
Association between bacterial/fungal infection between other complications of cirrhosis、organ failure、AKI or ACLF. | From admission to discharge, an average of 28-day
  Association between bacterial/fungal infection between other complications of cirrhosis、organ failure、AKI or ACLF.
Difference in type of organ failure between bacterial/fungal infection and other precipitating events. | From admission to discharge, an average of 28-day
  Difference in type of organ failure between bacterial/fungal infection and other precipitating events.
ACLF and each sub-type organ failure development at 28-day | From admission to discharge, an average of 28-day
  ACLF defined as per EASL CLIF-C or NACSELD definition Organ failure defined as per CLIF-C OF criteria, including Liver, coagulation, kidney, brain, respiratory and circulatory.
Transplantation-free Survival at 90-day | From admission to 90 day post-admission
  Survival at 90-day follow-up without liver transplantation
Overall survival at 28-、90-day | From admission to 90 day post-admission
  Overall survival at 28-、90-day
Readmission and further decompensations rate at 90-day post discharge | From admission to 90 day post-discharge
  Readmission and further decompensations rate at 90-day post discharge

CONTACTS AND LOCATIONS:
Overall Officials: Qing Xie, M.D., Ph.D., Principal Investigator — Ruijin Hospital
Locations (23):
- China (23):
  - First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Department of Critical Care Medicine of Liver Disease, Beijing You'an Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Department of severe Liver Diseases, Fuzhou Municipal Infectious Disease Hospital, Mengchao Hepatobiliary Hospital of Fujian Medical University,, Fuzhou, Fujian
  - Xiamen Hospital of Traditional Chinese Medicine, Xiamen, Fujian
  - Department of Infectious Disease, The First Hospital of Lanzhou University, Lanzhou, Gansu
  - The First People's Hospital of Lanzhou City, Lanzhou, Gansu
  - The Third People's Hospital of Guilin, Guilin, Guangxi
  - Department of Infectious Disease, The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Department of Infectious Diseases, Third Affiliated Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Department of Liver Diseases, The Third People's Hospital of Changzhou, Changzhou, Jiangsu
  - Department of Infectious Diseases, the Fifth People's Hospital of Suzhou, Suzhou, Jiangsu
  - The Fifth People's Hospital of Wuxi, Affiliated to Jiangnan University, Wuxi, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Department of Cirrhosis, Institute of Liver Disease, Shuguang Hospital, Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Department of Hepatology and Infection, Tongren Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Department of Infectious Diseases , Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Department of Infectious Diseases, First Affiliated Hospital of Xi'an Jiaotong University., Xi’an, Shanxi
  - Department of Infectious Diseases, Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The first Hospital of Jiaxing, Jiaxing, Zhejiang
  - Ningbo no.2 Hospital, Ningbo, Zhejiang
  - First Affiliated Hospital, Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No